CLINICAL TRIAL: NCT05019105
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Escalating Doses of ALKS 1140 With a Pilot Evaluation of Food Effect in Healthy Adult Subjects
Brief Title: Phase 1 ALKS 1140 in Healthy Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALKS 1140-001
Record Dates: First submitted 2021-08-16; First posted 2021-08-24 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Central Nervous System Diseases
MeSH Terms: conditions — Central Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo administered orally
  Interventions: Drug: Placebo
- ALKS 1140 (Active Comparator): Up to 8 single ascending doses of ALKS 1140 and 4 multiple ascending doses administered orally
  Interventions: Drug: ALKS 1140

INTERVENTIONS:
Drug: Placebo — Oral matching placebo
  Arms: Placebo
Drug: ALKS 1140 — Active oral dose of ALKS 1140
  Arms: ALKS 1140

SUMMARY:
To evaluate the safety and tolerability of ALKS 1140 in healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥18 and <30 kg/m2

Exclusion Criteria:

* Clinically significant illness or disease including significant cardiac, gastrointestinal (stomach)
* Subjects who have known allergic reactions to food or medications
* Women of childbearing potential
* Any clinically significant lifetime history of suicidal behavior or ideation (thoughts)
* Subject had lymphoma, leukemia, or any malignancy within the past 5 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Up to 28 days
Change in Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to 28 days
  Change in C-SSRS measured in Multiple-Ascending Dose subjects only
12-lead safety ECG results | Up to 28 days
  ECG parameters (Heart Rate, RR, PR, QRS, QT, QTcF, T wave) will be analysed using descriptive summary statistics (mean, standard deviation, median, minimum, and maximum for continuous variables) and as a change from baseline by dose level and treatment group. For the QT interval assessment, clinically abnormal ECG results for QTcF will be tabulated by protocol-specified millisecond range categories by dose and treatment group. Potentially clinically significant findings will be summarized by dose and treatment group.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) for ALKS 1140 | Measured at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 hours and Day 29
Time to Cmax (Tmax) | Measured at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 hours and Day 29
Half-life (t1/2) of ALKS 1140 | Measured at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours
Time until first quantifiable concentration (tlag) | Measured at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 hours and Day 29
Area under the concentration-time curve (AUC) | Measured at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 hours and Day 29
Apparent volume of distribution at terminal phase (Vz/F) | Measured at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 hours and Day 29
Apparent total clearance following oral administration (CL/F) | Measured at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and Day 29
Change from baseline in QTcF (Fridericia method) interval in response to treatment (Holter monitoring) | Measured at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and Day 29
Accumulation Index (RA) | Measured at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and Day 29

CONTACTS AND LOCATIONS:
Locations (1):
- Alkermes Clinical Investigative Site, Brisbane, Australia

IPD SHARING:
Plan to Share IPD: No